CLINICAL TRIAL: NCT04929691
Title: The CircumVent Project: A CPAP/O2 Helmet Solution for Non-Invasive Ventilation Using an Implementation Research Framework
Brief Title: The CircumVent Project: A CPAP/O2 Helmet Solution for Non-Invasive Ventilation Among Patients With COVID-19
Acronym: CircumVent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: New York University (Other)
Collaborators: Aliko Dangote Foundation (Unknown); Nigerian Institute of Medical Research (Other Government); CDC Foundation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDC Foundation Award 1085.1
Record Dates: First submitted 2021-06-08; First posted 2021-06-18 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: SARS-CoV-2 Acute Respiratory Disease; COVID-19 Respiratory Infection
Keywords: non-invasive ventilation; implementation science

STUDY DESIGN:
Intervention Model Description: The study will occur in 4 stages: 1) Convene a Steering Committee of key stakeholders and recruit implementation sites; 2) Use the integrated Promoting Action on Research Implementation in Health Services (i-PARiHS) framework to guide a needs assessment of treatment centers' capacity to use high-flow oxygen therapy to treat COVID-19 patients, and utilize the findings to develop an implementation strategy for use of CPAP/ O2 helmet solution; 3) Build infrastructure to support training and data monitoring processes and to develop implementation protocols to evaluate the adaptability of the strategy for the use of the CPAP/O2 helmet; and 4) Train health workers, distribute a CPAP/O2 helmet solution for non-invasive ventilation, pilot test the implementation strategy, and assess feasibility of its use and acceptability that includes monitoring altered risk of SARS-CoV-2 infection among healthcare workers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CPAP- Helmet Users (Experimental): Patients admitted to a study site with suspected or confirmed COVID-19 and who consented to using the CPAP helmet
  Interventions: Device: CPAP helmet
- Non-CPAP helmet users (Active Comparator): Patients admitted to a study site with suspected or confirmed COVID-19 but who did not use a CPAP helmet
  Interventions: Other: Standard of care non-helmet based CPAP ventilation

INTERVENTIONS:
Device: CPAP helmet — helmet-based CPAP ventilation for eligible patients; assess the feasibility and acceptability of the helmet-based CPAP ventilation
  Arms: CPAP- Helmet Users
Other: Standard of care non-helmet based CPAP ventilation — Standard of care ventilation without helmet-based CPAP
  Arms: Non-CPAP helmet users

SUMMARY:
The purpose of the CircumVent Project is to evaluate the feasibility, adaptability and acceptability of a CPAP/O2 helmet solution for non-invasive ventilation among patients with COVID-19 and health workers in eight COVID-19 treatment and isolation centers in Nigeria.

DETAILED DESCRIPTION:
Acute respiratory failure, a major cause of death in COVID-19, is managed with high-flow oxygen therapy via invasive mechanical ventilation. In resource-limited settings like Nigeria the shortage of ventilators and oxygen supply make this option challenging. Evidence-based non-invasive alternatives to mechanical ventilation such as the use of continuous positive airway pressure (CPAP) devices exist, but there have been concerns that non-invasive ventilation may expose healthcare workers to infection from aerosolized dispersion of SARS-CoV-2. The investigators propose to evaluate the feasibility, adaptability and acceptability of a CPAP/O2 helmet solution for non-invasive ventilation among patients with COVID-19 and health workers in eight COVID-19 treatment and isolation centers in Nigeria.

The study will occur in 4 stages: 1) Convene a Steering Committee of key stakeholders and recruit implementation sites; 2) Use the integrated Promoting Action on Research Implementation in Health Services (i-PARiHS) framework to guide a needs assessment of treatment centers' capacity to use high-flow oxygen therapy to treat COVID-19 patients, and utilize the findings to develop an implementation strategy for use of CPAP/ O2 helmet solution; 3) Build infrastructure to support training and data monitoring processes and to develop implementation protocols to evaluate the adaptability of the strategy for the use of the CPAP/O2 helmet; and 4) Train health workers, distribute a CPAP/O2 helmet solution for non-invasive ventilation, pilot test the implementation strategy, and assess feasibility of its use and acceptability that includes monitoring altered risk of SARS-CoV-2 infection among healthcare workers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to a study site with respiratory distress and suspected or confirmed COVID-19 infection

Exclusion Criteria:

* Patients who do not meet eligibility criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory rate | 1-4 weeks while on admission
  mild, 11-19/min; moderate, 20-24/min; severe, 25-30/min; very severe, >30 or <=10/min
Pulse Oximetry | 1-4 weeks while on admission
  mild >90; moderate <=90; severe, <88
Disposition | 1-4 weeks while on admission
  Died; Improved; Intubated

SECONDARY OUTCOMES:
Feasibility of using CPAP/O2 helmet solution | 1- 4 weeks while on admission
  Feasibility of Intervention Measure (FIM, Weiner et al. 2017), 4-item instrument with a 5-point ordinal scale (1 = minimum, 5 = maximum) that takes < 5 minutes to complete. Higher scores imply better outcome (greater feasibility).
Adaptability of the strategy for implementing CPAP/O2 helmet solution | 1-4 weeks while on admission
  Qualitative description of helmet use adaptations via self-report; Observed adaptation to patient characteristics
Acceptability of CPAP/O2 helmet solution for non-invasive management of COVID-19 | 1-4 weeks while on admission
  Acceptability of Intervention Measure (AIM, Weiner et al. 2017), a 4-item instrument with a 5-point ordinal scale (1= minimum, 5 = maximum). Higher scores imply better outcome (greater acceptability).

CONTACTS AND LOCATIONS:
Overall Officials: Babatunde L Salako, MBBS, FRCP, Study Director — Nigerian Institute for Medical Research, Lagos, Nigeria
Locations (9):
- Nigeria (9):
  - Nigerian Institute of Medical Research, Yaba, Lagos
  - Federal Medical Center, Abeokuta, Abeokuta
  - Alex Ekwueme Federal University Teaching Hospital, Enugu
  - Enugu State University Teaching Hospital, Enugu
  - University College Hospital, Ibadan
  - Aminu Kano Teaching Hospital, Kano
  - Federal Medical Center, Ebute Metta, Lagos
  - Lagos University Teaching Hospital, Lagos
  - Delta State University Teaching Hospital, Oghara

IPD SHARING:
Plan to Share IPD: No
Any study data to be shared will need to conform to Nigeria national data regulations.

REFERENCES:
- [Background] Patel BK, Wolfe KS, MacKenzie EL, Salem D, Esbrook CL, Pawlik AJ, Stulberg M, Kemple C, Teele M, Zeleny E, Macleod J, Pohlman AS, Hall JB, Kress JP. One-Year Outcomes in Patients With Acute Respiratory Distress Syndrome Enrolled in a Randomized Clinical Trial of Helmet Versus Facemask Noninvasive Ventilation. Crit Care Med. 2018 Jul;46(7):1078-1084. doi: 10.1097/CCM.0000000000003124. PMID 29595563
- [Background] Liu Q, Gao Y, Chen R, Cheng Z. Noninvasive ventilation with helmet versus control strategy in patients with acute respiratory failure: a systematic review and meta-analysis of controlled studies. Crit Care. 2016 Aug 23;20(1):265. doi: 10.1186/s13054-016-1449-4. PMID 27549178
- [Background] Beitler JR, Owens RL, Malhotra A. Unmasking a Role for Noninvasive Ventilation in Early Acute Respiratory Distress Syndrome. JAMA. 2016 Jun 14;315(22):2401-3. doi: 10.1001/jama.2016.5987. No abstract available. PMID 27179463
- [Background] Brambilla AM, Aliberti S, Prina E, Nicoli F, Del Forno M, Nava S, Ferrari G, Corradi F, Pelosi P, Bignamini A, Tarsia P, Cosentini R. Helmet CPAP vs. oxygen therapy in severe hypoxemic respiratory failure due to pneumonia. Intensive Care Med. 2014 Jul;40(7):942-9. doi: 10.1007/s00134-014-3325-5. Epub 2014 May 10. PMID 24817030
- [Background] Chiumello D, Brochard L, Marini JJ, Slutsky AS, Mancebo J, Ranieri VM, Thompson BT, Papazian L, Schultz MJ, Amato M, Gattinoni L, Mercat A, Pesenti A, Talmor D, Vincent JL. Respiratory support in patients with acute respiratory distress syndrome: an expert opinion. Crit Care. 2017 Sep 12;21(1):240. doi: 10.1186/s13054-017-1820-0. PMID 28899408
- [Background] Delclaux C, L'Her E, Alberti C, Mancebo J, Abroug F, Conti G, Guerin C, Schortgen F, Lefort Y, Antonelli M, Lepage E, Lemaire F, Brochard L. Treatment of acute hypoxemic nonhypercapnic respiratory insufficiency with continuous positive airway pressure delivered by a face mask: A randomized controlled trial. JAMA. 2000 Nov 8;284(18):2352-60. doi: 10.1001/jama.284.18.2352. PMID 11066186
- [Derived] Ahonkhai AA, Musa AZ, Fenton AA, Aliyu MH, Ofotokun I, Hornstein A, Musa BM, Nwosu N, Ulasi I, Ajayi S, Falade C, Dada A, Abdu A, Sunday M, Odewabi A, Rotimi MK, Ogueh O, Steinbach A, Ogedegbe G, Salako BL, Ezechi OC. The CircumVent Project: a CPAP/O2 helmet solution for non-invasive ventilation using an implementation research framework. Implement Sci Commun. 2021 Aug 26;2(1):93. doi: 10.1186/s43058-021-00193-y. PMID 34446110